CLINICAL TRIAL: NCT05967624
Title: Feasibility and Acceptability of a Low-cost, Mobile Telemedicine Platform for Remote Assessment of Children Transported by Ambulance
Brief Title: Prehospital Telemedicine Feasibility/Acceptability Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: H-38282; 5K23HL145126-03 (NIH)
Record Dates: First submitted 2023-07-21; First posted 2023-08-01 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Respiratory Distress Syndrome
Keywords: Teleconsultation
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Remote Consultation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Teleconsultation group (Experimental): Eligible children managed by urban paramedic teams responding to 911 calls in the prehospital setting to support a future trial of clinical efficacy.
  Interventions: Other: Teleconsultation

INTERVENTIONS:
Other: Teleconsultation — Each subject will be remotely assessed by a Medical Control Physician (MCP) using Zoom Pro (HIPAA-compliant video-conferencing software) on tablet devices as a low-cost mobile telemedicine platform and the Respiratory Observation Checklist, validated for telemedicine use in emergency settings. All prehospital clinical decision making will be made at the discretion of evaluating paramedics as per standard state-approved protocols and procedures, independent of checklist results.

SUMMARY:
Teleconsultation, or the use of video telecommunications technology to deliver expert recommendations for care remotely, has been used to improve the safety and quality of emergency care for children in hospital-based acute care settings by providing real-time access to remote pediatric physician experts. Whether extending teleconsultation as a patient safety intervention to emergency medical systems (EMS) outside hospitals can similarly benefit sick and injured children in the community is unknown. Advances in mobile technology have made teleconsultation more accessible and affordable for EMS systems. However, this intervention has been underutilized by EMS partially due to the lack of prehospital research supporting its efficacy for pediatric applications.

In prior simulation studies, the investigators found high intervention acceptance among key stakeholder groups (pediatric emergency physicians and paramedics), and demonstrated that it was feasible to integrate video communication into prehospital clinical workflows involving critical care delivery in high-risk pediatric scenarios. These initial simulation studies were conducted in a controlled prehospital setting in static ambulances using infant simulator manikins to minimize risk to children and providers. Demonstrating feasibility and acceptability with real children in moving ambulances is the next step to build the necessary evidence base to support future planned prehospital efficacy trials with children.

The investigators hypothesize that remote respiratory assessment of children by medical control physicians (expert physicians) using a mobile teleconsultation platform is acceptable to users (physicians and transport providers), and technically feasible in real transports.

DETAILED DESCRIPTION:
An open-label, nonrandomized, pilot feasibility trial will be conducted of children with respiratory distress transported by the Boston Children's Hospital (BCH) critical care transport team that also serves Boston Medical Center (BMC). Transport providers will initiate a video-call from the ambulance to medical control physician on call who will be at a geographically distant location. The physician will view streamed video of the child and complete a brief respiratory assessment checklist tool to determine video quality, a feasibility measure.

The investigators will measure acceptability (primary outcome) and feasibility (secondary outcomes) on a validated questionnaire administered to users after each call. In this pilot study, efficacy will not be tested; all decision making will occur according to usual care protocols.

ELIGIBILITY:
Inclusion Criteria:

* Children in New England transported by the Boston Children Hospital for respiratory illness from any cause
* Clinically stable for transportation [e.g., need supplemental oxygen, medications, or are stable on mechanical ventilation]

Exclusion Criteria:

* Children with non-respiratory complaints
* Children whose illness is anticipated by providers to be acutely life-threatening during transportation [e.g., requiring emergency resuscitation procedures in the ambulance]
* Non-English speaking parents/guardians

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2024-06-10 (Actual); Primary Completion 2025-02-14 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Agreement in assessment of respiratory distress | 6 months
  Each subject will be remotely assessed by a Medical Control Physician using the HIPAA-compliant Zoom Pro web application pre-loaded on a tablet device. The remote medical control physician and the transport team member at the patient bedside in the ambulance will score the Respiratory Observation Checklist simultaneously. The range for agreement is 0 to 1.0, where 0=no agreement and 1 is perfect agreement. The following scale: 0.01-0.20=none to slight, 0.21-0.40=fair, 0.41-0.60=moderate, 0.61-0.80=substantial, 0.81-1.0=almost perfect agreement will be used.

SECONDARY OUTCOMES:
Total Usability Score | 6 months
  The total usability score is measured by the Telehealth Usability Questionnaire (TUQ). This 21-item questionnaire is a validated measure of all the key usability characteristics of telehealth platforms (usefulness, ease of use, effectiveness, reliability, and satisfaction). Users rate items on 7-point Likert-scales (1=disagree to 7=agree) in 6 separate domains (usefulness, ease of use and learnability, interface quality, interaction quality, reliability, satisfaction and future use). The investigators modified this questionnaire to specifically address the usability of the study telemedicine platform. The total usability score is the total mean score for all 21 questions (maximum possible score=7).
Video quality | 6 months
  This will be measured by TUQ items #11 and #14 within the "Interaction Quality" domain. Users will rate each item on a 7-point Likert-scale (1=disagree to 7=agree), so scores will range from 1 to 7. The mean score and standard deviation (SD) for each item will be reported. HIgher scores suggest higher quality.
Audio quality | 6 months
  This will be measured by TUQ items #12 and #13 within the "Interaction Quality" domain. Users will rate each item on a 7-point Likert-scale (1=disagree to 7=agree), so scores will range from 1 to 7. The mean score and SD for each item will be reported. HIgher scores suggest higher quality.
Success of video-call connection | 6 months
  The number of attempts transport team providers make to successfully connect with the medical control physician via video-call will be recorded. Adequate success of video-call connection is defined as ≤2 attempts to achieve a video-call connection.
Proportion of successful tablet mounts | 6 months
  Study investigators will note any problems with tablet mounts in the ambulance cabin (e.g., location makes call activation difficult), as well as specific qualitative comments from participants regarding tablet mount strategy. If no problems are noted the tablet mount will be considered successful and the proportion of successful table mounts will be reported.
Proportion of calls with adequate video quality for assessment | 6 months
  This will be measured as the proportion of video-calls where clinicians are able to observe all ten items on the Respiratory Observation Checklist. This checklist tool has been previously validated for rapid, reliable assessment of children by teleconsultants in emergency settings. Medical control physicians will score 9 observable signs and a global assessment of respiratory distress dichotomously (present/absent).
Time to arrival at referring facility | 6 months
  This is the time interval (minutes) from when BCH receives the patient transport request from the referring facility to the time the transport team arrives at the referring facility. This will be abstracted from transport records.
Scene time | 6 months
  This is the time interval (minutes) from when the BCH transport team arrives at the referring facility to when the transport team leaves the referring facility. This will be abstracted from transport records.
Time to arrival at destination facility | 6 months
  This is the time interval (minutes) from when the BCH transport team leaves the referring facility to the time of arrival at BCH/BMC (the destination facility). This will be abstracted from transport records.
Total transport time | 6 months
  This time interval encompasses the time from when the transport team is dispatched to the referring facility to when they arrive at the destination (receiving facility). This will be abstracted from transport records.

CONTACTS AND LOCATIONS:
Overall Officials: Tehnaz Boyle, MD PhD, Principal Investigator — Boston Medical Center
Locations (2):
- United States (2):
  - Boston Children's Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-05-09): https://cdn.clinicaltrials.gov/large-docs/24/NCT05967624/ICF_000.pdf